CLINICAL TRIAL: NCT02443181
Title: The Application of DBS Technologies for Demand-driven Management of Essential Tremor
Brief Title: Demand-driven Management of Essential Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Andrew Ko, Assistant Professor, Department of Neurological Surgery, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00001079
Record Dates: First submitted 2015-04-28; First posted 2015-05-13 (Estimated); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Essential Tremor
Keywords: Essential tremor; closed-loop DBS
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Activa PC+S (Experimental): Patients will be implanted with standard DBS electrodes for treatment of essential tremor, at the Vim nucleus of the thalamus, and an additional subdural electrode array overlying hand motor cortex.. The patient will receive standard of care programming for thalamic stimulation for essential tremor. During research study visits, implementation and evaluation of closed-loop DBS using the PC+S system will be performed.
  Interventions: Device: Activa PC+S

INTERVENTIONS:
Device: Activa PC+S — Implementation of closed loop DBS for essential tremor

SUMMARY:
This study evaluates the effectiveness of tremor control using various strategies for implementing demand-driven thalamic deep brain stimulation (DBS) for essential tremor. Therapeutic stimulation at the Vim nucleus of the thalamus will be initiated and modulated using signals derived from external sensors (e.g. EMG, accelerometer) and cortical or thalamic electrodes.

DETAILED DESCRIPTION:
Essential tremor is effectively treated with deep brain stimulation of the ventralis intermedius nucleus of the thalamus, presumably because high-frequency stimulation disrupts aberrant cerebellar-thalamic input. For the most part, patients with essential tremor have a kinetic tremor that is present or worsened with movement. However, DBS therapy is currently continuous, and thus, stimulation occurs when the patient will not benefit symptomatically from treatment. This exposes the patient to unnecessary stimulation, which can lead to unnecessary usage of battery, unnecessary exposure to stimulation side-effects, and can possibly contribute to tolerance to DBS therapy.

One possible solution is selective stimulation when movement is required. This study will determine signals predictive of motor activity using external sensors such as EMG, and cortical biomarkers of real and imaginary movement that are well-characterized.

The primary aim is to demonstrate successful initiation and modulation of DBS therapy using the Activa PC+S system and implanted cortical or thalamic electrodes. Putative improvements in battery usage related to stimulation on-time and definition of coupling signals between thalamus and cortex that characterize tremor state are secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Appropriate candidates for DBS with essential tremor

Exclusion Criteria:

* Not meeting inclusion criteria based on tremor amplitude, neuropsychological testing, etc.
* Prior trauma to the brain on side of putative implantation of stimulator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-02; Primary Completion 2022-02 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 18 months
  Adverse events will be tracked using CTCAE terminology.

SECONDARY OUTCOMES:
Battery usage using demand-driven strategies for tremor control | 18 months
  Battery usage will be measured as stimulation on-time and voltage over time using demand-driven stimulation paradigms versus continuous stimulation paradigm.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ko, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Department of Neurological Surgery, Seattle, Washington, United States